CLINICAL TRIAL: NCT01190488
Title: Feasibility Of An Advanced Care Decision Aid Among Patients And Physicians
Brief Title: Feasibility Of An Advanced Care Decision Aid Among Patients And Physicians_Matlock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-0819; 630-92754 (Other Grant/Funding Number: Foundation for Informed Medical Decision Making); NCT01235611 (obsolete NCT alias)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Palliative Care; Decision Making; Decision Support Techniques; Decision Support Systems, Clinical; Hospices
Keywords: End of life decision making; End of life decision aid; Palliative care decision making; Palliative care decision aid; Advanced care planning; Decision Aid
MeSH Terms: interventions — Death Domain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - Decision Aid (Experimental): In addition to usual care, patients assigned to the intervention group will also be asked to view and/or read the EOL-PtDA during their hospitalization. The EOL-PtDA can be utilized anytime in the course of their hospitalization (all hospital rooms at UCH have a DVD player). This could be before, during, or after the palliative care team consultation.
  Interventions: Behavioral: End-of-Life / Advanced Care Decision Aid
- Active comparison (Active Comparator): Patients assigned to the control group will receive usual care which includes a discussion of knowledge about their medical condition as well as their goals of care. Typically, this discussion includes one physician and one advanced practice nurse however there are occasions such as weekends and during clinic time where the consult will have only one palliative care team member. This consultation typically includes a discussion of advanced directives using the five wishes document.
  Interventions: Behavioral: Active Comparator

INTERVENTIONS:
Behavioral: End-of-Life / Advanced Care Decision Aid — Patients assigned to the control group will receive usual care which includes a discussion of knowledge about their medical condition as well as their goals of care. Typically, this discussion includes one physician and one advanced practice nurse however there are occasions such as weekends and during clinic time where the consult will have only one palliative care team member. This consultation typically includes a discussion of advanced directives using the five wishes document.
  Other Names: FIMDM; Looking Ahead: Choices for medical care when you're seriously ill
  Arms: Intervention - Decision Aid
Behavioral: Active Comparator — TAU
  Arms: Active comparison

SUMMARY:
The investigators propose an evaluation of an end of life patient decision aid (EOL-PtDA) developed by the Foundation for Informed Medical Decision Making using the RE-AIM (Reach Effectiveness, Adoption, Implementation, and Maintenance) framework. To evaluate the Reach and Effectiveness, the investigators propose a pilot randomized clinical trial of the EOL-PtDA among patients on the inpatient palliative care service at University Hospital in Colorado. To evaluate barriers and facilitators of Adoption, Implementation, and Maintenance of the EOL-PtDA, we propose focus groups of non-palliative care physicians as we perceive these physicians to be the largest barrier to ultimate adoption of the EOL-PtDA. Additionally we propose a focus group of the palliative care physicians who participated in the implementation of this decision guide study to evaluate the feasibility of conducting a randomized control trial within a pall. care service and to evaluate the acceptability of this decision aid as it was implemented. The investigators also propose to conduct focus groups of normal, healthy clinic patients to determine the acceptability among that population. The End-of-Life decision aid is different from other decision aids. From the vantage point of decision quality, a major difference is that its primary focus is on helping patients clarify their values rather than gain knowledge. The results from this study will provide critical preliminary data to inform a randomized clinical trial and/or widespread implementation of the EOL-PtDA.

Specific Aims/Research question(s):Aim 1: To determine the Reach and Effectiveness of an end-of-life patient decision aid by conducting a pilot randomized clinical trial in an inpatient palliative care service. Aim 2: To determine physicians' attitudes towards the end-of-life patient decision aid and to gain insights into potential barriers and facilitators to Adoption, Implementation, and Maintenance by conducting a qualitative study of non-palliative care, and separately, palliative care physicians. Aim 3: To determine healthy clinic patients' attitudes towards the end-of-life patient decision aid and to gain insight into its Reach and Effectiveness.

DETAILED DESCRIPTION:
The aims 2-3 of this study include focus groups for physicians (both palliative care and non-palliative care physicians, aim 2) as well as healthy clinic patients (aim 3). Since these two arms are not randomized, they are not reported here. For additional information on the protocol and findings, please contact the PI, Daniel.Matlock@ucdenver.edu or the study coordinator, Tarah.Keech@ucdenver.edu.

ELIGIBILITY:
Inclusion Criteria:

* For Aim 1: To determine the Reach and Effectiveness of an end-of-life patient decision aid by conducting a pilot randomized clinical trial in an inpatient palliative care service.

Participants/Setting: Inpatient Palliative Care Service - University of Colorado Hospital: Patients may be included in this study if they are hospitalized at University of Colorado Hospital (UCH) and the UCH inpatient palliative care service has been consulted. This service, which consists of 6 physicians and two advanced practice nurses, sees approximately 40 new consults per month. More than 30% of consults originate from the hematology and oncology services, with the bulk of the remaining consults originating from the critical care services, cardiology, internal medicine, pulmonology and oncologic surgery. More than half of consults are for "goal clarification," others are for assistance with symptom control or disposition issues. We have chosen this population for the pilot because they are a high risk population with significant advanced care planning needs and they are captive and easily accessible to both PIs of this study. We will include adult patients and/or decision makers (ages 18 or greater) with end-of-life decisional needs as judged by the practitioners on the palliative care service. In cases where the patient is unable to participate due to an altered mental status, the person identified as the decision maker will be invited to participate in the study. Patients will be considered eligible if the UCH palliative care service has been consulted for "goal clarification" and/or assistance with end-of-life discussions rather than symptom control.

Exclusion Criteria:

* For Aim 1: We will exclude patients who cannot speak English or who are visually impaired as the decision aid is visual and only available in English. We will also exclude patients and decision makers with cognitive impairment as determined by ability to consent to the study. Ability to consent will be determined by the potential subject's ability, after being informed, to comprehend and explain the purposes, risks and benefits, and components of the study. If through the consent process, we determine that the person designated as the decision maker is unable to consent to the study, we will notify the primary team taking care of this patient. Additionally, we will exclude patients for whom the primary decision maker is unclear.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Healthcare trajectory | For intervention group, post intervention. For AC group, >= 24 hours after first assessment.
  We will follow enrolled patients for the duration of the study and examine the following metrics: days in the ICU, place of death, resuscitation status, chemotherapy, feeding tube, discharge disposition and re-hospitalization status. Patients in both groups will be asked to complete a brief quantitative survey.

SECONDARY OUTCOMES:
Quantitative measures of knowledge and values items | For intervention group, post intervention. For AC group, >= 24 hours after first assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Matlock, MD, MPH, Principal Investigator — UCD, UCH
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States